CLINICAL TRIAL: NCT05411705
Title: A Multicenter Randomized Controlled Study to Assess the Efficacy and Safety of rhTPO's Prophylactic Treatment of Cancer Treatment-induced Thrombocytopenia in Patients With High Risk of Treatment-induced Cardiac Injury
Brief Title: Efficacy and Safety of rhTPO's Prophylactic Treatment of CTIT in Patients With High Risk of Cardiac Injury
Acronym: Circular
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Anqing Municipal Hospital (Other); Henan Cancer Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Peking University Shougang Hospital (Other); Chinese PLA General Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Henan Provincial People's Hospital (Other); Shanxi Provincial Cancer Hospital (Unknown); Beijing Sanhuan Cancer Hospital (Unknown); Hebei Medical University Fourth Hospital (Other); Tongji Hospital (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Bethune Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Xia Yunlong, Director, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJ-KS-KY-2022-28(X)
Record Dates: First submitted 2022-05-26; First posted 2022-06-09 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Cancer Treatment Induced Thrombocytopenia
Keywords: rhTPO; Prophylactic Treatment; Cancer Treatment Induced Thrombocytopenia; Treatment Induced Cardiac Injury
MeSH Terms: interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTPO (Experimental): The study in a 2:1 randomization ratio (110 subjects to rhTPO).
  Interventions: Drug: rhTPO
- Control (Other): The study in a 2:1 randomization ratio (55 subjects to control group).
  Interventions: Drug: Control

INTERVENTIONS:
Drug: rhTPO — rhTPO 300U/kg/d QD, subcutaneous injection applied for 5 days per cycle, total 3 cycles. If the patient's platelet count showed a trend of continuous decline and/or was accompanied by the risk of bleeding during the treatment or after the completion of 5 doses of rhTPO, the investigator judged that rhTPO should be continued for treatment, and rhTPO could be administered subcutaneously at 300U/kg/ day for a maximum of 14 doses per cycle. Discontinue when the absolute platelet count increases by ≥50×10^9/L or when the platelet count rises to ≥250×10^9/L.
  Other Names: Recombinant human thrombopoietin; TPIAO
  Arms: rhTPO
Drug: Control — Non-rhTPO treatment
  Other Names: No intervention
  Arms: Control

SUMMARY:
To assess the efficacy and safety of an optimised dosing regimen of rhTPO's prophylactic treatment of cancer treatment-induced thrombocytopenia(CTIT) and to explore the cardioprotective effect of rhTPO in cancer patients with high risk of treatment-induced cardiac injury.

DETAILED DESCRIPTION:
This is an open-label prospective randomized multicenter study of rhTPO's prophylactic treatment of CTIT in patients receiving chemotherapy at high risk of cardiac injury. Adult cancer patients with high risk of cancer treatment-induced thrombocytopenia and cardiac injury were enrolled. Patients will be randomised into the rhTPO treatment group or non-rhTPO treatment group with a 2:1 ratio. The patients in rhTPO group will receive rhTPO 300U/kg/d subcutaneous injection for 5 days per cycle and total 3 cycles. The primary endpoint is to observe the improvement of platelet count by rhTPO during 3 cycles treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than or equal to 18 years of age at signing of the informed consent.
* Patients clinically judged to be at high risk of CTIT: Patients who had a platelet count below 50×10^9/L in the past 3 months; or patients who meet the criteria for prophylactic treatment in the Chinese Expert Consensus on the Management of Thrombocytopenia due to Oncology Chemotherapy (2018 Edition).The criteria for prophylactic treatment include: 1) The nadir platelet value in the last chemotherapy cycle was <50×10^9/L；Or 2)The patients with nadir platelet value ≥50×10^9/L and <75×10^9/L in the previous chemotherapy cycle also met at least one of the following risk factors for bleeding:

  1. With a previous history of bleeding.
  2. Chemotherapy regimens containing platinum, gemcitabine, cytarabine, anthracycline, etc.
  3. Combination regimens containing targeted or chemotherapy drugs which regularly result in thrombocytopenia.
  4. Thrombocytopenia caused by bone marrow infiltration of tumor cells.
  5. Eastern Cooperative Oncology Group (ECOG) score ≥2.
  6. Previous radiotherapy or ongoing radiotherapy, especially for long and flat bones (e.g. pelvis, sternum, etc.).
* Platelet count ≥75×10^9/L and <150×10^9/L, Hemoglobin ≥9.0 g/dL and absolute neutrophils ≥1.5×10^9 /L during screening.
* Patients with medium and high-risk with cardiotoxicity risk score (CRS) ≥3 and ECOG score of 0, 1, or 2 during screening.
* The current tumor treatment belongs to the scope of neoadjuvant, adjuvant, relapsed metastatic/advanced first-line and second-line therapies, anticipated to receive at least 2 cycles of current regimen with survival ≥ 6 months. The regimens may be 14-day, 21-day or 28-day cycles combined with targeted, immunotherapy, etc.
* Inclusion of organ tumours and lymphomas, with no restriction on the type and stage of organ tumours, etc.
* Patient provided signed informed consent

Exclusion Criteria:

* Patients with severe cerebrovascular disease (including but not limited to stroke, cerebrovascular accident, etc.) or serious heart disease (such as heart valve disease, arrhythmia, myocardial infarction, congenital heart disease, cardiomyopathy, heart failure, etc.) within the 3 months.
* Previous thrombocytopenia caused by non-oncology chemotherapy drugs within 6 months, including but not limited to primary immune thrombocytopenia, EDTA-dependent pseudo-thrombocytopenia, hypersplenism, etc.
* Patients with blood dysplasia-related diseases such as aplastic anemia, myeloproliferative diseases, multiple myeloma, myelodysplastic syndromes, etc.
* Patients with any arterial and venous thrombotic events within the past 6 months；
* Patients who had agents that increase platelet production or transfusion of platelets within the past 1 month.
* Abnormal liver function:

  * Patients without liver metastasis: ALT/AST > 3ULN (upper limit of normal value) and TBIL > 3ULN.
  * Patients with liver metastasis: ALT/AST≥5ULN, TBIL≥5ULN.
* Abnormal renal function: Scr≥1.5ULN or eGFR≤60ml/min.
* Patients with uncontrolled serious infection;
* Pregnant women or those planning to have children during the study period and breastfeeding patients.
* Any condition that the investigator considers inappropriate for inclusion in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients whose platelet count is ≥ 75×10^9/L after 2 cycles cancer treatment. | After 2 cycles cancer treatment (month 1.5~month 2, depends on chemotherapy regimen), each cycle is 14, 21 or 28 days
  Efficacy was defined as treatment without salvage therapy to increase platelet counts.

SECONDARY OUTCOMES:
Proportion of patients receiving salvage treatment to increase platelet counts. | during 3 cycles cancer treatment period(each cycle is 14, 21 or 28 days)
  Salvage treatment including platelet infusion, rhIL-11, etc.
Changes in cTnT/cTnI | 1 and 3 months after initial treatment
Changes in NT-proBNP | 1 and 3 months after initial treatment
Changes in LVEF | 1 and 3 months after initial treatment
  LVEF will be assessed by echocardiography
Changes in neutrophile granulocyte count | during 3 cycles cancer treatment period(each cycle is 14, 21 or 28 days)
Incidence of adverse events | from study start date to the end of follow-up, up to 3 months
  treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yunlong Xia, MD,PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (15):
- China (15):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chaoyang District Sanhuan Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Affiliated Tumor Hospital of Nantong University, Nanyang, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shaanxi Provincial Cancer Hospital, Xi'an, Shaanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP
Time Frame: From 12 months 36 months after study completion.
Access Criteria: Upon request to PI.